CLINICAL TRIAL: NCT01486407
Title: An Observational Study of Intubating Conditions Comparing Intraosseous Vascular Access With Peripheral Intravenous Access for Drug Delivery in Rapid Sequence Intubation
Brief Title: Observational Study of Rapid Sequence Intubation Drug Delivery Using Intraosseous and Intravenous Access.
Status: Terminated | Type: Observational
Why Stopped: For poor enrollment
Sponsor: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Organization: Teleflex (Industry)
Other Study IDs: 2011-13
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Airway Control
Keywords: Airway management

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intravenous (IV) drug delivery: patients on whom intravenous vascular access has been established for the purpose of rapid sequence intubation drug delivery.
- Intraosseous (IO) drug delivery: Patients on whom intraosseous vascular access has been established for rapid sequence intubation drug delivery.

SUMMARY:
This study will evaluate using intraosseous vascular access and intravenous vascular access to give patients the necessary medications to perform rapid sequence intubation, for patients with airway difficulties. The investigators think the device operator will find the intraosseous and intravenous routes equal for drug delivery.

DETAILED DESCRIPTION:
This observational study will evaluate the intubating conditions of patients receiving rapid sequence intubation when receiving paralytic drug delivery via intravenous or intraosseous vascular access from the perspective of the medical professional performing rapid sequence intubation. The investigators believe that medical professionals will find equal intubating conditions for intravenous and intraosseous drug delivery.

ELIGIBILITY:
Inclusion Criteria:

* Requires rapid sequence intubation
* Succinylcholine is chosen paralytic agent
* Intravenous (IV) or Intraosseous (IO) access has been established for rapid sequence intubation
* For IV access patients, their rapid sequence intubation case is the next occurring IV rapid sequence intubation case following an enrolled IO Rapid Sequence Intubation (RSI) case.

Exclusion Criteria:

* Vascular access other than IV or IO has been established

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the emergency department with airway difficulties requiring rapid sequence intubation.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen W Borron, MD, Principal Investigator — Texas Tech University Health Science Center
Locations (2):
- United States (2):
  - Christus Spohn Hospital Corpus Christi, Corpus Christi, Texas
  - Texas Tech University Health Science Center El Paso, El Paso, Texas

REFERENCES:
- [Background] Reades R, Studnek JR, Vandeventer S, Garrett J. Intraosseous versus intravenous vascular access during out-of-hospital cardiac arrest: a randomized controlled trial. Ann Emerg Med. 2011 Dec;58(6):509-16. doi: 10.1016/j.annemergmed.2011.07.020. PMID 21856044
- [Background] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Background] Leidel BA, Kirchhoff C, Bogner V, Braunstein V, Biberthaler P, Kanz KG. Comparison of intraosseous versus central venous vascular access in adults under resuscitation in the emergency department with inaccessible peripheral veins. Resuscitation. 2012 Jan;83(1):40-5. doi: 10.1016/j.resuscitation.2011.08.017. Epub 2011 Sep 3. PMID 21893125
- [Background] Deakin CD, Nolan JP, Sunde K, Koster RW. European Resuscitation Council Guidelines for Resuscitation 2010 Section 3. Electrical therapies: automated external defibrillators, defibrillation, cardioversion and pacing. Resuscitation. 2010 Oct;81(10):1293-304. doi: 10.1016/j.resuscitation.2010.08.008. No abstract available. PMID 20956050
- [Background] Kleinman ME, de Caen AR, Chameides L, Atkins DL, Berg RA, Berg MD, Bhanji F, Biarent D, Bingham R, Coovadia AH, Hazinski MF, Hickey RW, Nadkarni VM, Reis AG, Rodriguez-Nunez A, Tibballs J, Zaritsky AL, Zideman D; Pediatric Basic and Advanced Life Support Chapter Collaborators. Pediatric basic and advanced life support: 2010 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendations. Pediatrics. 2010 Nov;126(5):e1261-318. doi: 10.1542/peds.2010-2972A. Epub 2010 Oct 18. No abstract available. PMID 20956433
- [Background] Brierley J, Carcillo JA, Choong K, Cornell T, Decaen A, Deymann A, Doctor A, Davis A, Duff J, Dugas MA, Duncan A, Evans B, Feldman J, Felmet K, Fisher G, Frankel L, Jeffries H, Greenwald B, Gutierrez J, Hall M, Han YY, Hanson J, Hazelzet J, Hernan L, Kiff J, Kissoon N, Kon A, Irazuzta J, Lin J, Lorts A, Mariscalco M, Mehta R, Nadel S, Nguyen T, Nicholson C, Peters M, Okhuysen-Cawley R, Poulton T, Relves M, Rodriguez A, Rozenfeld R, Schnitzler E, Shanley T, Kache S, Skippen P, Torres A, von Dessauer B, Weingarten J, Yeh T, Zaritsky A, Stojadinovic B, Zimmerman J, Zuckerberg A. Clinical practice parameters for hemodynamic support of pediatric and neonatal septic shock: 2007 update from the American College of Critical Care Medicine. Crit Care Med. 2009 Feb;37(2):666-88. doi: 10.1097/CCM.0b013e31819323c6. PMID 19325359
- [Background] Von Hoff DD, Kuhn JG, Burris HA 3rd, Miller LJ. Does intraosseous equal intravenous? A pharmacokinetic study. Am J Emerg Med. 2008 Jan;26(1):31-8. doi: 10.1016/j.ajem.2007.03.024. PMID 18082778
- [Background] Orlowski JP, Porembka DT, Gallagher JM, Lockrem JD, VanLente F. Comparison study of intraosseous, central intravenous, and peripheral intravenous infusions of emergency drugs. Am J Dis Child. 1990 Jan;144(1):112-7. doi: 10.1001/archpedi.1990.02150250124049. PMID 1688484
- [Background] Laurin EG, Sakles JC, Panacek EA, Rantapaa AA, Redd J. A comparison of succinylcholine and rocuronium for rapid-sequence intubation of emergency department patients. Acad Emerg Med. 2000 Dec;7(12):1362-9. doi: 10.1111/j.1553-2712.2000.tb00493.x. PMID 11099426
- [Background] Perry JJ, Lee JS, Sillberg VA, Wells GA. Rocuronium versus succinylcholine for rapid sequence induction intubation. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD002788. doi: 10.1002/14651858.CD002788.pub2. PMID 18425883

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous (IV) Drug Delivery | Intraosseous (IO) Drug Delivery
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous (IV) Drug Delivery | Intraosseous (IO) Drug Delivery | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (6.36) | 41 (56.57) | 40.25 (32.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time From First Drug Delivery to Operator-perceived Sufficient Relaxation to Perform Endotracheal Tube Placement
Description: Time measured in seconds from first drug delivery to the time of operator-perceived sufficient relaxation to perform endotracheal tube placement
Time Frame: during rapid sequence intubation procedure, average expected time frame 30 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intravenous (IV) Drug Delivery | Intraosseous (IO) Drug Delivery
Number analyzed (Participants) | 2 | 2
seconds | 62.5 (2.12) | 45 (21.21)

2. Primary Outcome: Intubation Difficulty Scale
Description: Intubation Difficulty Scale (IDS) provides a numerical Total score describing the difficulty of the intubation procedure based upon the summation of the following individual sub-scores:
  number of attempts (each additional attempt adds (+)1 point, minimum score=0, no maximum), number of operators (each additional +1 point, minimum score=0, no maximum), use of alternative techniques (each alternative technique +1 point, minimum score=0, no maximum), cormack grade for first oral attempt (measures the quality of the view of the larynx using grades 1 - 4 where higher number means poorer visibility; successful blind intubation=0. minimum score=0, maximum=4), lifting force required (normal=0 or increased=1), laryngeal pressure (not applied=0 or applied=1), vocal cord mobility (abduction=0 or adduction=1).
  Total IDS minimum score=0, no maximum score. Score 0=Easy; Score 1 - 5 =slight difficulty; Score >5 =moderate to major difficulty Score infinite =Failed/Impossible intubation
Time Frame: during rapid sequence intubation procedure, average expected time frame 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous (IV) Drug Delivery | Intraosseous (IO) Drug Delivery
Number analyzed (Participants) | 2 | 2
units on a scale | 1.5 (0.71) | 2 (1.41)

3. Primary Outcome: Operator Satisfaction With Intubating Conditions Using Visual Analog Scale
Description: Operator reported level of satisfaction with intubating conditions regarding adequacy of sedation and adequacy of muscular relaxation. This is reported using a 100 mm visual analog scale from 0 - 100 where higher numbers indicate greater satisfaction.
Time Frame: during rapid sequence intubation procedure, average expected time frame 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous (IV) Drug Delivery | Intraosseous (IO) Drug Delivery
Number analyzed (Participants) | 2 | 2
units on a scale | 95.75 (6.01) | 92.25 (0.35)

4. Primary Outcome: Failure Rate of Endotracheal Intubation and Requirement for Alternative Airway Management Methods
Description: Failure rate of endotracheal intubation and requirement for alternative airway management methods
Time Frame: during rapid sequence intubation procedure, average time frame 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous (IV) Drug Delivery | Intraosseous (IO) Drug Delivery
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

5. Secondary Outcome: Incidence of Short-term Catheter Related Complications for Each Technique
Description: Incidence of short-term catheter related complications for each technique (IO vs IV)
Time Frame: during emergency department stay, average time frame 24 hours
Measure: Number; unit: complications
Arm/Group | Intravenous (IV) Drug Delivery | Intraosseous (IO) Drug Delivery
Number analyzed (Participants) | 2 | 2
complications | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of participants stay in the Emergency Department, up to 24 hours.
Description: In this observational study only adverse events (AEs) associated with the IV or IO vascular access catheter(s) used during the rapid sequence intubation procedure were collected.
Arm/Group | Intravenous (IV) Drug Delivery | Intraosseous (IO) Drug Delivery
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less